CLINICAL TRIAL: NCT01842854
Title: Validation of Galectin-3 as a Biomarker for Determining Patients Prognosis With Chagas Disease
Brief Title: Galectin-3 as a Biomarker in Patients With Chagas Disease
Status: Completed | Type: Observational
Sponsor: Hospital Sao Rafael (Other)
Responsible Party: Principal Investigator, Milena Botelho Pereira Soares, PhD, Hospital Sao Rafael
Other Study IDs: CEP-41-10; Galectin-Chagas (Registry Identifier: CEP HSR 41-10)
Record Dates: First submitted 2013-04-18; First posted 2013-04-30 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Chagas Disease
Keywords: Galectin-3; Chagas disease; Biomarkers
MeSH Terms: conditions — Chagas Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, Serum, Whole Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Chagas disease diagnosis: Diagnosis of Chagas disease in both forms: indeterminate and cardiac ones, with and without ventricular dysfunction.

SUMMARY:
The purpose of this study is to analyze the efficacy of Galectin-3 as a biomarker on the Chagas Disease prognosis. This analysis will be done through the correlation between the plasmatic levels of this molecule with functional and laboratory tests.

DETAILED DESCRIPTION:
Previous studies indicate that activated macrophages secrete Galectin-3, a molecule that is involved in the development of fibrosis and tissue rearrangement in the liver, kidney and the heart. Its plasmatic levels are increased on patients with acute decompensated heart failure. These observations suggest that measuring levels of Galectin-3 in patients with cardiac diseases can be useful to determine their prognosis. To investigate the role of this new biomarker in Chagas Disease, we will study a Chagas Disease population (including patients with the indeterminate and cardiac form of the disease). The assessment of the prognostic value of Galectin-3 will be done through the comparison between its plasmatic levels and each patients's clinical evaluation, disease severity, inflammatory biomarkers and cardiac function tests.

The patients included in the study must at first sign the written consent. They shall be accompanied in the specialized outpatient clinics for Chagas disease - Hospital São Rafael - Centro de Biotecnologia e Terapia Celular. They will be submitted to several tests, including:

* Collection of Blood samples for biochemical analysis;
* Electrocardiogram;
* Holter Electrocardiogram;
* Echocardiogram;
* Treadmill Test;
* X-Ray Imaging;
* Magnetic Resonance Imaging;
* Evaluation of the quality of life through the application of questionnaires (SF 36 and the Minnesota Living With Heart Failure Questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* Chagas Disease diagnosis confirmed by 2 different serologies
* Diagnosis of indeterminate form or cardiac form, with and without ventricular dysfunction.

Exclusion Criteria:

* Significant valve disease defined as aortic stenosis with a gradient of VE/Ao > 50 mmHg
* Mitral stenosis with a valve area inferior than 1,5 cm2
* Severe or moderate aortic and/or mitral regurgitation
* Chronic use of immunosuppressive agents
* Dialysis treatment of terminal renal failure
* Fever on the last 48 hours or evidence of systemic infection in activity according to the definition of sepsis of the ACCP/SCCM (American College os Chest Physicians/Society of Critical Care Medicine)
* Current abusive use of alcohol or illicit drugs (Based on the DSM IV)
* Any other comorbidities that impact patient's survival within the next 2 years
* Liver disease in activity
* Continuous use of steroids as treatment for COPD
* Hematologic, neoplastic or bone diseases
* Homeostasis disturbances
* Inflammatory diseases or chronic infectious diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary Hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Correlation of plasmatic levels of Galectin-3 with the percentage of heart fibrosis | One year
  Mensuration of heart fibrosis percentage with Magnetic Resonance Imaging

SECONDARY OUTCOMES:
Correlation of plasmatic levels of Galectin-3 with the functional capacity of the heart | One year
  Mensuration of the functional capacity with treadmill test
Correlation of plasmatic levels of Galectin-3 with the serum levels of Pro-BNP. | One year
Correlation of plasmatic levels of Galectin-3 with the serum levels of TNF-alpha | One year
Correlation of plasmatic levels of Galectin-3 with the serum levels of IFN-gamma. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Milena Botelho Pereira Soares, PhD, Principal Investigator — Hospital São Rafael; Ricardo Ribeiro dos Santos, MD, PhD, Study Director — Hospital São Rafael; Ticiana Ferreira Larocca, MD, MSC, Study Chair — Hospital São Rafael; Márcia Maria Noya Rabelo, MD, MSC, Study Chair — Hospital São Rafael; Luís Cláudio Lemos Correia, MD, PhD, Study Chair — Hospital São Rafael; Bruno Solano de Freitas Souza, MD, MSC, Study Chair — Hospital São Rafael; Carolina Thé Macedo, MD, Study Chair — Hospital São Rafael
Locations (1):
- Hospital São Rafael, Salvador, Estado de Bahia, Brazil

REFERENCES:
- [Derived] Noya-Rabelo MM, Larocca TF, Macedo CT, Torreao JA, Souza BS, Vasconcelos JF, Souza LE, Silva AM, Ribeiro Dos Santos R, Correia LC, Soares MB. Evaluation of Galectin-3 as a Novel Biomarker for Chagas Cardiomyopathy. Cardiology. 2017;136(1):33-39. doi: 10.1159/000447529. Epub 2016 Aug 23. PMID 27548475